CLINICAL TRIAL: NCT04651907
Title: Efficacy of Acupuncture on Chemotherapy-Induced Peripheral Neuropathy (CIPN): A Phase III, Randomized, Sham-controlled Clinical Trial
Brief Title: Efficacy of Acupuncture on Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH109-REC3-121
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Keywords: acupuncture; chemotherapy-induced peripheral neuropathy; neuropathic pain; von-Frey monofilament test; taxane; platinum
MeSH Terms: conditions — Neuralgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture group (Experimental): The needle set for the sham acupuncture group and the real acupuncture group will use the CASOON Acupuncture Needle (Wuxi Jiajian Medical Instrument Company, limited), which needle size is 0.3mm×30mm. The needle placed for the real acupuncture group will be the same needle size as 0.3mm×30mm. The depth of needling varied based on the patient's body sizes. After insertion, the needles were manually manipulated to obtain the De Qi sensation, which was defined as the acupuncturist feeling a tugging or grasping sensation from the needle manipulation and the patient feeling soreness, fullness, heaviness, or local distension at local needling sites.
  Interventions: Other: acupuncture
- sham-controlled group (Placebo Comparator): The sham acupuncture group will be performed by superficial needling with less than 4mm depth. The needling location is about 0.5 cm away from the acupoints. Both the real acupuncture group and the sham acupuncture group received the same treatment protocol.
  Interventions: Other: minimal acupuncture
- waitlist-controlled group (No Intervention): As an waitlist control group, no acupuncture will be performed.

INTERVENTIONS:
Other: acupuncture — use disposable sterile steel needles to insert to the acupuncture point
  Arms: acupuncture group
Other: minimal acupuncture — The sham-controlled group will be performed with minimal acupuncture (superficial needling) at non-acupoints.
  Arms: sham-controlled group

SUMMARY:
The purpose of this study is to assess the neurological efficacy of acupuncture in patients with cancer who experienced peripheral neuropathy, which is induced by chemotherapy.

DETAILED DESCRIPTION:
Background: Chemotherapy may lead to peripheral neuropathy up to 40% in cancer survivors, especially in some types of patients with cancer. The effect of acupuncture, an ancient Chinese medicine technique, was recognized by the World Health Organization (WHO) in the treatment of several diseases. The postulated mechanisms associated with acupuncture in analgesia or neurogenesis are still under investigation. Considering a moderate recommendation for duloxetine in the treatment of chemotherapy-induced peripheral neuropathy (CIPN) based on based on neuropathic pain, and a few treatment options with evidence for CIPN, acupuncture might be another option. Nowadays, only small scale pilot studies provided initial proof of acupuncture in CIPN, particularly in decreasing neuropathic pain and improving neurotoxicity, the study aims to determine the beneficial effects of acupuncture on CIPN with a large-scale, multicenter, randomized sham-controlled clinical trial. Furthermore, the aim of the study will provide evidence for the clinical therapeutic guideline of CIPN in the future.

Methods: This three-armed, multicenter, randomized, parallel, sham-controlled clinical trial will conduct in three centers in Taiwan. We will randomly assign 234 eligible patients into three groups, an acupuncture group (n=90), a sham-controlled group (n=90), and a waitlist-controlled group (n=54). Each subject maintains the regular treatments of cancer except the chemotherapeutic agents designed in our design. The acupuncture group and the sham-controlled group will receive three therapeutic sessions each week for four weeks, and another two sessions each week for four weeks (a total of 20 sessions at eight weeks). Each group will be followed-up for four weeks, to evaluate the persistent efficacy of acupuncture. The sham-controlled group will be performed with minimal acupuncture (superficial needling) at non-acupoints. The primary outcome measurement will be the changes in the FACT-Ntx subscale from baseline to 20th acupuncture sessions. The secondary outcome will be the changes in BPI-SF average pain score from baseline to 20th acupuncture sessions. The third outcome will be the changes of target forces by von-Frey filament test at each point in hands and feet from baseline to 20th acupuncture treatments. from baseline to 20th sessions. FACT-Ntx scale and BPI-SF average pain score will be measured at four time-points, including baseline, the end of the 12th treatments, the end of the 20th treatments, and the end of the study at the 12th week. The von-Frey filament test will be measured at three-time points, including baseline, the end of the 20th treatments, and the end of the study at the 12th week.

ELIGIBILITY:
Inclusion Criteria:

The study will enroll patients with a symptom of peripheral neuropathy, including paresthesia, numbness, glove-and-stocking sensory loss distribution or pain in four limbs, and meet the following inclusion criteria:

1. All adult cancer patients (Age≧20-year-old) who received chemotherapy regimens, including adjuvant and neoadjuvant therapy
2. Stage I-III cancer patients
3. Completed chemotherapy regimens more than3 months, including Taxanes (paclitaxel or docetaxel), platinum (cisplatin, oxaliplatin, carboplatin)
4. Baseline von Frey Monofilament test (Target force at hand) ≧ 0.07gms
5. Baseline von Frey Monofilament test (Target force at foot) ≧ 0.4gms
6. Eastern Cooperative Oncology Group (ECOG) performance status ≦3
7. Grading of peripheral sensory neuropathy in National Cancer Institute- common terminology criteria for adverse events,v5.0 (NCI-CTCAE5) ≧1
8. Patients were restricted acupuncture treatment for one month before recruitment
9. Written patient informed consent

Exclusion Criteria:

Participants with any of the following conditions will be excluded:

1. Uncontrolled Diabetic Mellitus, HbA1c≧7% is inappropriate[19].
2. Diabetic neuropathy diagnosed before receiving chemotherapy
3. Neuropathy from any type of nerve compression (e.g., carpal/tarsal tunnel syndrome, radiculopathy, spinal stenosis, brachial plexopathy)
4. Concomitant with duloxetine, or another analgesia, including Pregabalin, Venlafaxine, Minocycline, Topical gel, Oxycodone, Naloxone, Cannabinoids, and Angiotensin II type 2 receptor antagonist
5. Severe hemorrhagic coagulopathy or bleeding tendency
6. Unstable cardiovascular disease
7. Severe skin lesions around the treatment sites The researchers will exclude any participants considered to be inappropriate for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of FACT-Neurotoxicity subscale(NtxS) | It will be assessed before the first session, after the 12th session, the 20th session, and followed at the end of the 12th week.
  The primary outcome will be the change FACT-Neurotoxicity subscale(NtxS) from baseline to 20 sessions at 8th weeks. The neurotoxicity subscale from the FACT/GOG-NTX-13(version 4) contains 13 items assessing numbness, tingling, and discomfort in the hands or feet, difficulty hearing, tinnitus, joint pain or muscle cramps, weakness, or trouble walking, buttoning buttons, or feeling small shapes when placed in the hand. Items are scored from 0-4 (0 = not at all; 4 = very much) and summed (total score range = 0-52). Since no published data are defining a cut-point for determining a clinically important change in the FACT/GOG Ntx score, we defined a 4 point change as a clinically meaningful improvement in patient-reported CIPN-related neurotoxicity outcome. The authorized translated traditional Chinese version will be purchased in this study.

SECONDARY OUTCOMES:
The change of BPI-SF | It will be assessed before the first session, after the 12th session, the 20th session, and followed at the end of the 12th week.
  Our secondary outcome will be the change of average pain severity in BPI-SF from baseline to 20 sessions at 8th weeks. BPI-SF is an instrument used to evaluate the severity of pain, including neuropathic pain and the interference on the patients' daily functioning. Items are scored from 0 to 10 (0= no pain; 10= pain as bad as you can imagine). Since not all the patients feel pain in their daily life, we selected the participants who have average pain severity more than 4 points at baseline assessment into the final analysis. The authorized translated traditional Chinese version will be purchased in this study.
The quantitative sensation of touch detection | It will be assessed before the first session, the 20th session, and followed at the end of the 12th week.
  The quantitative sensation of touch detection was used to test sensory levels and obtain objective data on the status of diminishing or returning sensibility. Touch detection was measured using von Frey monofilaments (Semmes-Weinstein Von Frey Aesthesiometer, Stoelting Co. 620 Wheat Lane, Wood Dale, IL, USA), with weights from 0.008 g to 300 g at 8 points. The measuring sites including the bases of the sole, tips of the big toe, palmar sides of hands, and the fingertips of the middle finger.The well-known up-down method applied to measure touch-detection thresholds.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hung Chen, Ph.D., Study Director — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No